CLINICAL TRIAL: NCT03083249
Title: Gardasil Anonymous Survey
Brief Title: Gardasil Knowledge
Status: Completed | Type: Observational
Sponsor: Sarah Hostetter, MD (Other)
Responsible Party: Sponsor-Investigator, Sarah Hostetter, MD, Principal Investigator, St. Louis University
Organization: St. Louis University (Other)
Other Study IDs: 27816
Record Dates: First submitted 2017-03-03; First posted 2017-03-17 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: HPV
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gardasil — None-data gathering only

SUMMARY:
Human papillomavirus (HPV) is the most common viral genital tract infection. The majority of women and men who are sexually active will be exposed to a strain or strains of the virus. While there are hundreds of viral strains, high risk strains are associated cervical and oral cancers. According to the Centers for Disease Control (CDC), between 2008 and 2012 there were 38,793 deaths attributed to HPV related cancers. Vaccinations were created in an attempt to prevent infection from the most common high risks strains of HPV. Gardasil/HPV-9 was created to help prevent HPV related cancers and warts. The HPV-9 vaccine includes protection from 7 strains of HPV associated with 74% of HPV related cancers. While Gardasil was approved and released in 2006, many men and women have not been vaccinated. A national immunization survey in 2011 of teens 13-17 years old noted that only 60% of girls and 40% of boys have received at least one vaccination in the series. While complete vaccination series is recommended, a recent study found that a single dose of Gardasil when compared to placebo created a higher level of serum antibodies in uninfected females.

DETAILED DESCRIPTION:
All patients seen at a single clinic will be offered participation in the anonymous survey. The survey will ask a series of questions regarding basic demographics, sexual history, smoking status, and Gardasil vaccine knowledge. The survey will serve as evidence of the vaccine utility by highlighting patient risk factors for HPV and patient knowledge about the vaccine series.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18-26 will be offered participation

Exclusion Criteria:

* Not meeting the inclusion criteria

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Females age 18-26 of all ethnic background
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
knowledge about HPV risk factors | 1 year
  The survey asks about Gardasil vaccine knowledge

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hostetter, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No